CLINICAL TRIAL: NCT05618418
Title: BActeriophages To Treat Liver Disease Eliminating Harmful Bacteria (BATTLE)
Acronym: BATTLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Frederik Cold, Principal Investigator, MD, Ph.d., Specialist Registrar in Medical Gastroenterology, Copenhagen University Hospital, Hvidovre
Other Study IDs: H-21041462
Record Dates: First submitted 2022-11-03; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Alcoholic Hepatitis
Keywords: Gut microbiome
MeSH Terms: conditions — Hepatitis, Alcoholic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Fecal samples collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospital admitted patients with alcoholic hepatitis: Inclusion criteria:
  Age ≥ 18 Bilirubin > 50 micromol/L History of large alcoholic consumption in period prior to hospital admission (in the last six months) No bile-duct obstruction (investigated through US, CT og MRI)
  Exclusion criteria:
  Hepatocellulary carcinoma Viral hepatitis Autoimmune hepatitis Portal thrombosis Pregnancy Expected survival for less than one year caused by other diseases (based on decision from project responsible doctors)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Alcoholic hepatitis is a disease with a high mortality rate with few treatment options improving survival. Recently certain bacterial strains has been correlated to survival in patients with alcoholic hepatitis.

In the BATTLE-trial the investigators will investigate if certain bacteria are correlated to decreased chance of survival in patients with alcoholic hepatitis.

DETAILED DESCRIPTION:
Patients with alcoholic hepatitis who are admitted to Copenhagen University Hospital Hvidovre and Herlev will be invited to participate.

Blood and fecal samples following hospital admission will be collected. Through one-year follow-up correlation of certain bacteria in fecal samples with survival will be investigated.

In particular whether patients with cytolysin producing E. faecalis has a decreased chance of survival compared to patients without this bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Bilirubin > 50 micromol/L
* History of large alcoholic consumption in period prior to hospital admission (in the last six months)
* No bile-duct obstruction (investigated through US, CT og MRI)

Exclusion Criteria:

* Hepatocellulary carcinoma
* Viral hepatitis
* Autoimmune hepatitis
* Portal vein thrombosis
* Pregnancy
* Expected survival for less than one year caused by other diseases (based on decision from project responsible doctors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital admitted patients with alcoholic hepatitis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Survival in patients with and without cytolysin producing E. faecalis in fecal samples | 6 months
  Patient alive/not alive - Cytolysin producing E. faecalis in fecal samples from hospital admission (yes/no)

SECONDARY OUTCOMES:
Survival in patients with and without cytolysin producing E. faecalis in fecal samples | 1 year
  Patient alive/not alive - Cytolysin producing E. faecalis in fecal samples from hospital admission (yes/no)
Survival in patients with and without cytolysin producing E. faecalis in fecal samples | 30 days
  Patient alive/not alive - Cytolysin producing E. faecalis in fecal samples from hospital admission (yes/no)
Survival in patients with and without cytolysin producing E. faecalis in fecal samples | 90 days
  Patient alive/not alive - Cytolysin producing E. faecalis in fecal samples from hospital admission (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: frederik cold, MD, PHD, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No
No plan to make data available to researchers